CLINICAL TRIAL: NCT01222325
Title: Comparison Between Two Shock Wave Regimens Using Frequencies of 60 and 90 Impulses Per Minute for Urinary Stones
Brief Title: Comparison Between Two Shock Wave Regimens for Treating Urinary Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: EDUARDO MAZZUCCHI, University of Sao paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1183/06
Record Dates: First submitted 2010-10-05; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2009-08

CONDITIONS: Urinary (Renal or Ureteral) Stones
Keywords: kidney calculi; urolithiasis; urologic surgical procedures; extracorporeal shockwave lithotripsy
MeSH Terms: conditions — Calculi; Kidney Calculi; Urolithiasis | interventions — Lithotripsy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- swl 3000 impulses- 60 imp/min (Active Comparator): patients in this group were submitted to extracorporeal shockwave lithotripsy (SWL) 3000 impulses at 60 impulses per minute under general anesthesia. Unique session
  Interventions: Procedure: extracorporeal shockwave lithotripsy (SWL)
- swl- 4000 impulses - 90 impulses /min (Active Comparator): patients in this group were submitted extracorporeal shockwave lithotripsy (swl) to 4000 impulses at 90 impulses per minute under general anesthesia- unique session
  Interventions: Procedure: extracorporeal shockwave lithotripsy (SWL)

INTERVENTIONS:
Procedure: extracorporeal shockwave lithotripsy (SWL) — patients were submitted to one session SWL at a Dornier Compact Delta lithotripter under general anesthesia under supervision of an anesthesiologist and an urologist.
  Other Names: lithotripsy; shock waves

SUMMARY:
In order to check if a reduction in the frequency and total number of shocks delivered during extracorporeal shockwave lithotripsy (SWL) results in a great number of stone-free patients,the investigators compared two different ways of treating urinary stones using SWL.

DETAILED DESCRIPTION:
Purpose: Two different regimens of SWL delivery for treating urinary stones were compared.

Methods: After informed consent, patients with previously untreated renal and ureteric stones were admitted for an initial treatment by SWL between June 2008 and May 2009. Patients were randomly divided into two groups; one group received 3000 impulses at a rate of 60 impulses per minute, and the other received 4000 impulses at a rate of 90 impulses per minute. Patients submitted to re-treatment of the same stone were excluded. All treatments were done using the Dornier Compact Delta lithotripter. Stones were located by x-ray or ultrasound. Prior to treatment, patients were submitted to laboratory tests and a cardiologic evaluation when indicated. Urinary infections were treated prior to the SWL session. All procedures were performed under general anesthesia. Briefly, Tramadol 1-2 mg/kg associated to Propofol 2.5-3.0 mg/kg and scopolamine were employed in the majority of the procedures. Patients received 50-100 mg of diluted Tramadol and 20 mg of scopolamine just before the beginning of the SWL session and Propofol was maintained on continuous bomb infusion during the treatment and interrupted three minutes before the end of the session. All patients were maintained under spontaneous breathing, and a facial or a laryngeal oxygen mask was used according to the anesthesiologist's judgment. The potency of the lithotripter was increased progressively by 300 shocks until reaching the final stage, which occurred at a mean of 1500 shocks. The maximum potency employed was level 4 (equivalent to 14 kV) for renal stones and level 6 (16 kV) for ureteric stones.

All patients were treated on an outpatient basis and were discharged from the hospital six hours after treatment. All patients received non-steroidal anti-inflammatory drugs (NSAIDs) and Dipyrone in combination with to Hyoscine for three days postoperatively unless contraindicated and were instructed to come to the emergency department in case of severe pain, fever or hematuria.

The final results for each patient were assessed with a kidney and urinary bladder scan (KUB) plus an abdominal ultrasound three months after the procedure. Success was defined as stone-free status or the detection of residual fragments ≤ 3 mm on final evaluation. Partial fragmentation was considered to have occurred if a significant reduction in the stone burden was observed but residual fragments bigger than 3 mm remained.

We evaluated overall stone-free rates, the incidence of unchanged stones and the occurrence of partial fragmentation as well as the occurrence of significant complications in both groups.

The sample size required was based on the assumption that the estimated success rate would be 70% in the 3000 impulses at 60 impulses per minute group and 50% in the 4000 impulses at 90 impulses per minute group, with a type I error of 0.05 and a type II error of 0.05 (power of 80%). This yielded a projected sample size of 93 stones in each group.

Data were analyzed using the Fischer's exact, Chi-square and Mann-Whitney tests; a level of significance of 5% was adopted.

ELIGIBILITY:
Inclusion Criteria:

* patients with renal or ureteral stones from 5 to 20 mm

Exclusion Criteria:

* pregnancy
* coagulation disturbs and antiplatelet treatment
* urinary tract infection
* aortic aneurism bigger than 2 cm
* clinical contraindication to general anesthesia
* refusal in participating of the protocol

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
abdominal ultrasound and abdominal x rays (KUB) | 3 months
  patients submitted to SWL in two different regimens were submited to renal ultrasound and abdominal x rays (KUB) three months after procedure to check the occourrence of stone-free status, residual fragments or unmodified stone.

SECONDARY OUTCOMES:
adverse effects of the two different regimens | 3 months
  patients submitted to two different SWL regimens were followed clinically and submited to renal ultrasound and abdominal x ray to check the occurrence of adverse effects like hematoma or peri renal collections.

CONTACTS AND LOCATIONS:
Overall Officials: eduardo mazzucchi, md, Principal Investigator — univesrity of sao paulo general hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil